CLINICAL TRIAL: NCT00210951
Title: An Active Safety Surveillance Plan to Conduct Serologic Testing for Anti-erythropoietin Antibodies and Prospectively Monitor the Incidence of Pure Red Cell Aplasia (PRCA) Among Patients Receiving Epoetin Alfa or Another Erythropoietin
Brief Title: Study to Monitor the Incidence of Pure Red Cell Aplasia (PRCA) and/or Antibodies to Erythropoietin Among Participants Receiving Epoetin Alfa or Another Erythropoietin
Status: Completed | Type: Observational
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Other Study IDs: CR003925; EPO-IMU-402 (Other: Johnson & Johnson Pharmaceutical Research & Development, L.L.C.)
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Red-Cell Aplasia, Pure; Chronic Renal Failure
Keywords: Epoetin alfa; Erythropoietin; Red Cell Aplasia, Pure; Chronic Renal Failure
MeSH Terms: conditions — Red-Cell Aplasia, Pure; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Participants Receiving Epoetin Alfa or Another Erythropoietin: Participants will not receive any intervention in this study. Participants with chronic renal disease receiving treatment with epoetin alfa or other recombinant erythropoietins will be prospectively observed to monitor incidence of pure red cell aplasia and/or antibodies to erythropoietin. Participants will receive standard-of-care treatment for their chronic renal (or other) disease from their individual Investigators.
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — Participants will not receive any intervention in this study. Participants with chronic renal disease receiving treatment with epoetin alfa or other recombinant erythropoietins will be prospectively observed to monitor incidence of pure red cell aplasia and/or antibodies to erythropoietin. Participants will receive standard-of-care treatment for their chronic renal (or other) disease from their individual Investigators.

SUMMARY:
The purpose of this study is to assess the incidence of pure red cell aplasia (PRCA [suppression of erythropoiesis with little or no abnormality of leukocyte or platelet production]) among participants with chronic renal failure (CRF), who were receiving treatment with epoetin alfa or other exogenous recombinant erythropoietin therapies.

DETAILED DESCRIPTION:
This is a prospective (observation of a population for a sufficient number of persons over a sufficient number of years to generate incidence or mortality rates subsequent to the selection of the study group), observational (clinical study in which participants may receive diagnostic, therapeutic, or other types of interventions, but the investigator does not assign participants to specific interventions) and cohort study. Study specific information will be collected from participants with chronic renal disease who are receiving recombinant erythropoietin and their treatment course will be followed for up to 2 years and participants will not receive any intervention in this study. Upon entering the study, information will be collected regarding disease history and recombinant erythropoietin treatment. Every 3 months thereafter, progress information will be collected, including recombinant erythropoietin treatment, number of red blood cells and presence of any signs of pure red cell aplasia (PRCA) development. Blood samples will be collected at study entry and every 3 months. Participants discontinuing erythropoietin will be followed only for an additional 12 months from the time erythropoietin is discontinued. Participants will receive standard-of-care treatment for their chronic renal disease from their individual Investigators. Participants will be primarily observed prospectively for PRCA.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants of legal age to give consent according to local standards
* Participants must be receiving or about to receive treatment with an erythropoietin as part of a pre-existing treatment plan for their chronic renal (or other) disease
* Physicians treating the participants must agree in advance to document any appearance of pure red cell aplasia (PRCA) such that information and details of the case may be reported to regulatory agencies (with patient identification protected)
* If required by local ethics committees, participants must give consent to permit the collection of de-identified personal data for the specific purpose of this study and to collect blood samples for tests for antibodies to erythropoietin

Exclusion Criteria:

* Participants who are unable to complete future follow-up visits
* Participants who when entering the study have any of the following symptoms of pure red cell aplasia (PRCA): Loss of effectiveness of erythropoietin or low number of immature red blood cells while on erythropoietin as shown by a blood test or bone marrow examination
* Participants with a history of PRCA or loss of effectiveness with erythropoietin at the time of enrollment into the study
* Participants whose anemia did not respond to previous treatment with an erythropoietin
* Participants with a history of antibodies to erythropoietin prior to entering the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with chronic renal disease receiving treatment with epoetin alfa or other recombinant erythropoietins.
Sampling Method: Non-Probability Sample
Enrollment: 4761 (Actual)
Dates: Start 2003-05; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Pure Red Cell Aplasia (PRCA) | Up to 2 years
  The PRCA is the suppression of erythropoiesis with little or no abnormality of leukocyte or platelet production.
Number of Participants With Positive Serum Erythropoietin (EPO) Antibodies | Up to 2 years
  Antibodies are immunoglobulin molecules having a specific amino acid sequence by virtue of which they interact only with the antigen (or a very similar shape) that induced their synthesis in cells of the lymphoid series.
Relationship between EPO Antibodies and PRCA | Up to 2 years
  Natural history of EPO antibodies will be examined and its relationship to PRCA will be checked.

SECONDARY OUTCOMES:
Number of Participants With Pure Red Cell Aplasia (PRCA) Associated With Different Routes of Administration | Every 3 Months up to up to 2 years
  The PRCA is the suppression of erythropoiesis with little or no abnormality of leukocyte or platelet production.
Change From Baseline in Number of Participants With PRCA Over Time | Baseline and Month 3, 6, 9, 12, 15, 18, 21, 24
  The PRCA is the suppression of erythropoiesis with little or no abnormality of leukocyte or platelet production.
Duration of Exposure | Up to 2 years
  Duration of exposure to study medication is the time between the first and last dose of study medication.

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: An Active Safety Surveillance Plan to Conduct Serologic Testing for Anti-Erythropoietin Antibodies and Prospectively Monitor the Incidence of Pure Red Cell Aplasia (PRCA) Among Patients Receiving Epoetin Alfa or Another Erythropoietin — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=543&filename=CR003925_CSR.pdf